CLINICAL TRIAL: NCT05618444
Title: Enhancing Positive Positive Airway Pressure (PAP) Adherence Among Spanish-Speaking Hispanic Adults With Obstructive Sleep Apnea (OSA)
Brief Title: Enhancing PAP Adherence Among Spanish-speaking Hispanic Adults With OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0810
Record Dates: First submitted 2022-11-03; First posted 2022-11-16 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: positive airway pressure (PAP); adherence; Hispanic; tele-management
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated Management (AM) (Experimental): Receipt of text-based behavioral intervention
  Interventions: Behavioral: Automated Management (AM)
- Usual Care (No Intervention): Control group receiving usual care for obstructive sleep apnea

INTERVENTIONS:
Behavioral: Automated Management (AM) — A tele-management intervention that will deliver two-way messages to participants via a bot - a computer program that simulates human activity. Programmed AM messages will address evidence based intervention components for positive airway pressure (PAP) adherence, including PAP use awareness (tele-monitoring), support and troubleshooting, education, and brief motivational messaging.
  Arms: Automated Management (AM)

SUMMARY:
This study seeks to enhance long-term positive airway pressure (PAP) adherence among Spanish-speaking Hispanics, a group with known PAP outcomes disparities. This study will assess the feasibility of a linguistically and culturally adapted tele-management intervention (Automated Management, AM) for Spanish-speaking Hispanic adults with OSA.

DETAILED DESCRIPTION:
This feasibility study seeks to enhance long-term positive airway pressure (PAP) adherence among Spanish-speaking Hispanics, a group with known PAP outcomes disparities. This study will assess the feasibility, usability and 6-month effectiveness of a linguistically and culturally adapted efficacious tele-management intervention (Automated Management, AM) for Spanish-speaking Hispanic adults with obstructive sleep apnea (OSA) (N=50). A prospective, randomized, parallel group, unblinded, feasibility trial is proposed. AM is a tele-management strategy that includes evidence-based components for improving shorter-term PAP adherence consisting of education, support and troubleshooting, and brief targeted motivational enhancement delivered by tele-messaging. The automated two-way, interactive communication is algorithmic based on PAP use and behavioral profiles defined at baseline. The innovative, technology-based interventions are designed to ensure access to sustained care that overcomes barriers such as distance/geography, transportation limitations or lost work/productivity time. As such, AM can provide equitable access to quality long-term PAP management that may mitigate known PAP adherence disparities for minority adults with OSA. If effective for long-term PAP adherence, these strategies may alter OSA care paradigms, improve outcomes and associated healthcare costs, and reduce disparities.

ELIGIBILITY:
Inclusion Criteria:

* Spanish-speaking and reading
* Self-identified Hispanic
* Adults ≥ 18 years-old
* Males and females
* Moderate-severe OSA defined as AHI ≥15 events/hour using a hypopnea criterion of a 4% oxygen desaturation (AHI4%)
* Expected availability for the duration of the study (6 months from date of randomization)
* Ownership of smartphone with unlimited text messaging capability
* Referred to PAP treatment and able and willing to be treated with PAP

Exclusion Criteria:

* Other sleep apnea or nocturnal respiratory insufficiency or failure diagnosis other than OSA established by polysomnogram (PSG) or home sleep apnea test (HSAT)
* Requirement of supplemental oxygen or other non-invasive ventilation modality
* Women referred to PAP because of new-onset OSA with pregnancy as PAP treatment may be time-limited (enrolled women who become pregnant during the trial and are already on PAP treatment will not be excluded)
* Anticipated or scheduled bariatric surgery and/or referred to sleep evaluation by bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 6 months
  Satisfaction with quality of care and the components of care (e.g., feedback, frequency, duration), relevance of the care to the individual and their needs, and overall satisfaction with care. Assessed with the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 scores range from 8 to 32, with higher values indicating higher satisfaction.
Acceptability | 6 months
  Defined as the perception that a given treatment is agreeable, palatable, or satisfactory. Assessed with the Acceptability of Intervention Measure (AIM; 4 items, Likert, 1-5, where 1 = "completely disagree" and 5 = "completely agree"). Higher scores indicate higher acceptability.
Appropriateness | 6 months
  Defined as the perceived fit, relevance, or compatibility of a given treatment. Assessed with the Intervention Appropriateness Measure (IAM; 4 items, Likert, 1-5, where 1 = "completely disagree" and 5 = "completely agree"). Higher scores indicate higher appropriateness.

SECONDARY OUTCOMES:
Recruitment Rate | 6 months
  Recruitment Rate computed at the end of the trial
Retention Rate | 6 months
  Retention Rate computed at the end of the trial

OTHER OUTCOMES:
Positive airway pressure (PAP) use from 3-6 months | 3-6 months
  Hours of PAP use per 24 hours
PAP adherence based on modified Centers for Medicare & Medicaid Services (CMS) criteria | 6 months
  Adherence yes/no using ≥4 hours/night and ≥70% of nights
Patient Satisfaction | 1 month
  Satisfaction with quality of care and the components of care (e.g., feedback, frequency, duration), relevance of the care to the individual and their needs, and overall satisfaction with care. Assessed with the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 scores range from 8 to 32, with higher values indicating higher satisfaction.
Patient Satisfaction | 3 months
  Satisfaction with quality of care and the components of care (e.g., feedback, frequency, duration), relevance of the care to the individual and their needs, and overall satisfaction with care. Assessed with the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 scores range from 8 to 32, with higher values indicating higher satisfaction.
Acceptability | 1 month
  Defined as the perception that a given treatment is agreeable, palatable, or satisfactory. Assessed with the Acceptability of Intervention Measure (AIM; 4 items, Likert, 1-5, where 1 = "completely disagree" and 5 = "completely agree"). Higher scores indicate higher acceptability.
Acceptability | 3 months
  Defined as the perception that a given treatment is agreeable, palatable, or satisfactory. Assessed with the Acceptability of Intervention Measure (AIM; 4 items, Likert, 1-5, where 1 = "completely disagree" and 5 = "completely agree"). Higher scores indicate higher acceptability.
Appropriateness | 1 month
  Defined as the perceived fit, relevance, or compatibility of a given treatment. Assessed with the Intervention Appropriateness Measure (IAM; 4 items, Likert, 1-5, where 1 = "completely disagree" and 5 = "completely agree"). Higher scores indicate higher appropriateness.
Appropriateness | 3 months
  Defined as the perceived fit, relevance, or compatibility of a given treatment. Assessed with the Intervention Appropriateness Measure (IAM; 4 items, Likert, 1-5, where 1 = "completely disagree" and 5 = "completely agree"). Higher scores indicate higher appropriateness.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Saconi, PhD, Principal Investigator — Geisinger Clinic
Locations (4):
- United States (4):
  - Kaiser Permanent Southern California, Fontana, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Geisinger, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No